CLINICAL TRIAL: NCT00581698
Title: Intraoperative Mapping of Regional Lymphatics Draining the Primary Site of Melanoma Using Isosulfan Blue
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Daniel Coit, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 91-015
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Melanoma
Keywords: Melanoma; Negative regional lymph nodes; Primary melanomas Clark III and Breslow thickness > 1 mm, or Clark; IV-V and any Breslow thickness, and clinically negative regional nodes
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue (lymph node)

GROUPS / COHORTS (1):
- Surgical: Patients with primary melanomas Clark III and Breslow thickness > 1 mm, or Clark IV-V and any Breslow thickness, and clinically negative regional nodes

SUMMARY:
The purpose of this study is to determine whether we can consistently identify the first lymph node (the "sentinel node") draining your melanoma.

DETAILED DESCRIPTION:
The issue of elective lymph node dissection (LND) in the management of melanoma patients with clinically negative nodes remains controversial. The concept of elective LND is attractive because it provides the opportunity to detect and remove occult micrometastases before they become clinically apparent. Numerous retrospective analyses have consistently shown a 15-20% long term survival advantage in patients undergoing elective LND who are found to have positive nodes, compared to those undergoing therapeutic LND for clinically positive nodes. The majority of patients undergoing elective LND however, do not have lymph node involvement, and the impact of removal of these negative nodes on the survival of these patients is unknown. The substantial morbidity of these procedures has led to the conduct of a number of important prospective randomized trials designed to define the impact of elective LND on the survival of patients with clinically node negative melanoma. In 1982, the World Health Organization reported on the end results of 553

The primary objective of this protocol is to establish the feasibility of lymph node mapping, using preoperative lymphoscintigraphy and intraoperative blue dye injection to detect the sentinel node in patients at risk for regional lymph node metastasis from their primary melanoma.

ELIGIBILITY:
Inclusion Criteria:

* primary melanomas Clark III and Breslow thickness > 1 mm, or Clark IV-V and any Breslow thickness
* clinically negative regional nodes

Exclusion Criteria:

* previous definitive wide local excision of the primary melanoma with skin graft
* an inflammatory lesion in the area of the primary melanoma that is likely to drain to the same nodal basin
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary melanomas Clark III and Breslow thickness > 1 mm, or Clark IV-V and any Breslow thickness, and clinically negative regional nodes. Patients with a resectable solitary intransit metastasis and clinically negative nodes will be considered for entry on to this protocol on an individual basis.
Sampling Method: Non-Probability Sample
Enrollment: 876 (Actual)
Dates: Start 1991-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
This is a trial to assess the feasibility of the technique of identifying the sentinel node using the technique of lymphatic mapping as described by Morton. The primary endpoint of the trial will be success or failure in identifying the sentinel node. | 18 years 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Coit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org